CLINICAL TRIAL: NCT03396770
Title: Impact of the Early Hemodynamic Evaluation Guided by Urinary Biomarkers on the Acute Kidney Injury After Cardiac Surgery
Brief Title: Acute Kidney Injury After Cardiac Surgery
Acronym: NEPHROCAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: JRAR Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 35RC17_8822; 2017-A01935-48 (Other: ID-RCB)
Record Dates: First submitted 2017-12-15; First posted 2018-01-11 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Acute Kidney Injury; Cardiac Surgery
Keywords: Urinary biomarkers; Intensive Care Unit
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: open labeled randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Standard clinical routine
  Interventions: Procedure: Standard clinical routine
- Nephrocheck group (Experimental): Nephrocheck test
  Interventions: Procedure: Nephrocheck test

INTERVENTIONS:
Procedure: Standard clinical routine — Patient management is carried out according to the usual service protocol
  Arms: Control group
Procedure: Nephrocheck test — Nephrocheck® test is realized 4 hours after the end of the cardiopulmonary bypass
  * If the test is positive, hemodynamic evaluation is carried out and adapted therapy to result of this evaluation is initiated.
  * If the test is negative, patient management is carried out according to the usual protocol.
  * A second test is realized 6 hours after the first test whatever the result of it.
  Arms: Nephrocheck group

SUMMARY:
Acute kidney injury (AKI) is common after cardiac surgery. The diagnosis is based on the criteria defined by the Kidney Disease Improving Global Outcomes (KDIGO) classification: oliguria and elevation of serum creatinine. However, oliguria is not specific of AKI and elevation of serum creatinine is too late. Therefore, new methods have been developed to earlier assess the risk of AKI.

Among those methods, it has been shown that the increase of urinary dosage, in the hours following the surgery, of two proteins (Tissue Inhibitor of Metallo-Protease 2 (TIMP2) and Insulin Growth Factor Binding Protein 7 (IGFBP7)) is associated with an increased risk of occurrence of AKI in patients hospitalized in intensive care unit. The Nephrocheck® test combines the urinary dosage of those two proteins TIMP2 and IGFBP7.

Insofar as post-surgery low cardiac output is one curable cause of AKI, the early detection of early kidney risk allows corrective measures to stabilize hemodynamic state and thus to reduce the risk of AKI.

DETAILED DESCRIPTION:
The usual diagnostic markers of AKI are defaulted. Indeed, oliguria tends to overstate the impact of AKI, up to 40-50% of patients. Postoperative increased serum creatinine is a late marker for the AKI. Furthermore, perioperative hemodilution and serum creatinine kinetic delay the postoperative peak of serum creatinine from 48 to 72 h.

Nephrocheck® test combines the urinary dosage of 2 proteins (TIMP2 and IGFBP7). These 2 proteins are excreted by the tubular cell in case of suffering whatever the origin, for example tissue hypoxia by low renal blood flow or a systemic inflammatory response. In a medical ICU, the test performed within 4 to 12 hours after kidney aggression can predict the onset of persistent AKI beyond 4 weeks.

Until randomization, all patients are treated according to the standard of care for the center. This includes a blood test upon arrival in the intensive care unit and continuous monitoring of vital parameters.

ELIGIBILITY:
Inclusion Criteria:

* On-pump cardiac surgery ;
* Informed and written consent of the patient or inclusion according to the emergency procedure;
* Affiliated patient or beneficiary of a social protection

Exclusion criteria:

* Left and / or right ventricular assist device;
* Heart transplant;
* Chronic kidney disease with renal replacement therapy before surgery;
* Hemorrhagic shock requiring surgical hemostasis at the time of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 848 (Actual)
Dates: Start 2018-01-14 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Occurence of an AKI according to the KDIGO classification without oliguria | 72 hours after surgery
  According to the KDIGO classification:
  Stage 1; Increase in serum creatinine ≥ 26.5 μmol / l or 1.5 to 1.9 times baseline serum creatinine Stage 2; Increase in baseline serum creatinine from 2.0 to 2.9 times Stage 3; An increase of 3.0 times the baseline serum creatinine or serum creatinine ≥ 354 μmol / l or initiation of renal replacement therapy

SECONDARY OUTCOMES:
Filling solute volumes | 48 hours after surgery
  Recording of the filling solute volumes administered within 48 hours postoperatively
Use of catecholamin | 48 hours after surgery
  Recording (YES/NO) of the recourse of catecholamin required during the medical care, within 48 hours postoperatively
Special extra corporeal circulation | 48 hours after surgery
  Recording (YES/NO) of the recourse of a particular extracorporeal system within 48 hours postoperatively : Extracorporeal Life Support, heart pumps (Impela® like devices), or Intra-aortic balloon pump.
Duration of stay in the ward | Up to 28 days post surgery
Oliguria | 48 hours after surgery
  Proportion of patients with an oliguria defined according to the KDIGO criteria :
  * Stade 1 ; diuresis < 0.5 mL/kg/h for 6 à 12 h
  * Stade 2 ; diuresis < 0.5 mL/kg/h for more than 12h
  * Stade 3 ; diuresis < 0.3 mL/kg/h for more than 24h or anuria ≥ 12h ;
Repeatability of the Nephrocheck® test | 10 hours post surgery
  Only for the patients in the Nephrocheck arm, variations between pre and postoperative Nephrocheck® test results will be assessed
Mortality rate | Up to 28 days post surgery
  Mortality rate in the ward

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien BIEDERMANN, MD, Principal Investigator — CHU Rennes
Locations (1):
- Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: No